CLINICAL TRIAL: NCT01080274
Title: Vitamin D and Zinc Levels in Patients Undergoing Ergometry Test
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Renana Shor MD, Assaf-Harofeh Medical Center
Other Study IDs: 22/10
Record Dates: First submitted 2010-03-03; First posted 2010-03-04 (Estimated); Last update posted 2010-04-07 (Estimated); Status verified 2010-02

CONDITIONS: Atherosclerosis
Keywords: ergometry; vitamin d; zinc
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood will be collected for vit d and zinc , stored until all samples are collected and only than the laboratoty will analyze it.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- positive ergometry: positive ergometry as specified by a cardiologist on site.
- negative ergometry.: negative ergometry as specified by cardiologist on site.
- patients with positive stress test: 100 patients with positive ergometry test as specified by the cardiologist in charge. All patients are ambulatory patients referred for routine check up.

SUMMARY:
Low vitamin D levels were found to be associated with cardiovascular morbidity and mortality. Low zinc levels are associated with an increased atherosclerotic burden. Therefore we hypothesized that patients with pathological stress test would have low levels of Vitamin D and zinc compared to patients with a normal stress test.

DETAILED DESCRIPTION:
Hypovitaminosis D is generally defined as 25(OH)D levels of < 20ng/ml, while levels of 21-29ng/ml indicate insufficiency and those above 30ng/ml are regarded as sufficient.

The rational behind the observations associating vitamin D deficiency with CVD is that on the one hand, hypovitaminosis D was found to be associated with traditional risk factors such as hypertension (HTN),diabetes mellitus (dm),obesity, dyslipidemia and metabolic syndrome , on the other hand, experimental data demonstrated that vitamin D could affect cardiac muscle cells directly, control parathyroid (PTH) hormone secretion, regulate the rennin- angiotensin- aldosterone system and the immune system, all of which could influence cardiovascular risk.

Epidemiological studies further support this association, demonstrating high prevalence of hypovitaminosis D among U.S. adults with cardiovascular disease (74%). An association between low vitamin D levels and increased myocardial infarction risk as well as total mortality has been also observed.

Low 25hydroxyvitamin D[ 25(OH)D] levels were also independently associated with all cause and CVD mortality among patients scheduled for coronary catheterization.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* CCT > 60 ml/min
* No IHD
* No hyper/hypoparathyroidism
* No active malignancy
* Not taking calcium, phosphate

Exclusion Criteria:

* Under 18 years of age
* Not fulfilling inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Over 18 years old
  * CCT > 60 ml/min
  * No IHD
  * No hyper/hypoparathyroidism
  * No active malignancy
  * Not taking calcium, phosphate
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-03 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
positive stress test | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Assaf Harofeh Mc, Ẕerifin, Israel